CLINICAL TRIAL: NCT05241444
Title: Phase 1 Study of Autologous CD4^LVFOXP3 in Participants With Immune Dysregulation Polyendocrinopathy Enteropathy X-linked (IPEX) Syndrome
Brief Title: CD4^LVFOXP3 in Participants With IPEX
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bacchetta, Rosa, MD (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Jessie L. Alexander, Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-63373; DRU-2020-7764 (Other: FDA Office of Orphan Products Development); RPD-2020-470 (Other: FDA Office of Orphan Products Development); 1R01FD007540-01 (FDA); CLIN2-13259 (Other Grant/Funding Number: California Institute of Regenerative Medicine (CIRM))
Record Dates: First submitted 2022-01-12; First posted 2022-02-15 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: IPEX
Keywords: Treg cells; Regulatory T cells; Gene therapy; autoimmunity; Immune Dysregulation Polyendocrinopathy Enteropathy X-linked; FOXP3; Lentiviral; CD271; NGFR; immune suppression
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Escalating doses of CD4^LVFOXP3 will be administered in 2-6 participants per dose in two age cohorts (Cohort A: ≥ 12 years of age; Cohort B: < 12 years of age) using a 2+4 dose escalation design. Cohort B will be started at the second dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (≥12 years) (Experimental): The first participant in Dose Level 1 will be administered 1.0 x 10^6 CD4^LVFOXP3 /kg (± 20%).
  If there is no toxicity observed in the first participant, the following participants in Dose Level 1 will be administered the same dose of 1.0 x 10^6 CD4^LVFOXP3 /kg (± 20%).
  If there is no toxicity observed in any participants in Dose Level 1, participants will be enrolled into Dose Level 2 and administered 3 x 10^6 CD4^LVFOXP3 /kg (± 20%).
  If there is no toxicity observed in any participants in Dose Level 2, participants will be enrolled into Dose Level 3 and administered 10 x 10^6 CD4^LVFOXP3 /kg (± 20%).
  If in any dose level 1 of 2 participants show toxicity, that dose level will be expanded to 6 participants.
  Interventions: Biological: CD4^LVFOXP3
- Cohort B (<12 years) (Experimental): Participants in Cohort B will always follow treatment of participants in Cohort A for the same dose level.
  Cohort B will start at Dose Level 2 and be administered 3 x 10^6 CD4^LVFOXP3 /kg (± 20%).
  If there is no toxicity observed in any participants in Dose Level 2, participants will be enrolled into Dose Level 3 and administered 10 x 10^6 CD4^LVFOXP3 /kg (± 20%).
  If in any dose level 1 of 2 participants show toxicity, that dose level will be expanded to 6 participants.
  Interventions: Biological: CD4^LVFOXP3

INTERVENTIONS:
Biological: CD4^LVFOXP3 — Infusion of autologous CD4+ T cells that have undergone lentiviral-mediated gene transfer of:
  i) healthy human FOXP3 gene leading to persistent high FOXP3 expression and acquisition of Treg-like cell function; and ii) human CD271 surface marker gene that allows tracking and quantification of the CD4^LVFOXP3 in the blood.
  Other Names: CD4^LVFOXP3 Treg-like cells

SUMMARY:
This first-in-human, Phase 1 clinical trial will test the feasibility of the manufacturing and the safety of the administration of CD4^LVFOXP3 in up to 30 evaluable human participants with IPEX and evaluate the impact of the CD4^LVFOXP3 infusion on the disease.

DETAILED DESCRIPTION:
Treatment with CD4^LVFOXP3 is expected to replace the defective Treg cells of the participants, and restore control of the immune system and therefore ameliorate symptoms of IPEX.

We expect to learn the following from this study:

1. That CD4^LVFOXP3 can be consistently produced and be of expected quality to be used in humans,
2. That CD4^LVFOXP3 are safe in children and young adults with IPEX, and determine its effects, both good and bad,
3. That CD4^LVFOXP3 can improve overall health and allow reduction of medication/s.

This Phase 1 (feasibility and safety) trial will gather data about CD4^LVFOXP3 in vivo persistency and early signs of impact on symptoms of IPEX.

ELIGIBILITY:
Inclusion Criteria:

* Body weight greater than 8 kg, unless assessed as able to tolerate leukapheresis
* FOXP3 gene mutation
* Medical history of progressive symptoms of IPEX with persistency of some symptoms and/or signs requiring immune suppressive medication. The participant may or may not be on immunosuppression at time of starting the study.
* Uncontrolled IPEX disease but unable to tolerate immune suppressive medication
* Recurrent IPEX symptoms, requiring immune suppressive medications, in participants who have had prior allogeneic (allo) blood stem cell transplantation (HSCT).
* ≥ 50% Performance rating on Lansky/Karnofsky Scale
* Organ and marrow function within acceptable levels of function
* Absence of ongoing infections
* Must be able to consent if an adult

Exclusion Criteria:

* Medical instability
* Less than 6 months life expectancy
* Inability to meet limits for steroid dosing
* Eligible for an HLA matched sibling or matched unrelated donor blood stem cell transplant, and be willing to undergo transplant.
* Unrelated or comorbid disease
* Allergy to any study medication, product, or intervention
* Currently receiving another experimental treatment
* History of malignancy, unless disease free for at least 2 years, with the exception of non melanoma skin cancer or carcinoma in situ

Ages: 4 Months to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2037-02 (Estimated)

PRIMARY OUTCOMES:
Meet target cell number for dose manufacturing | Time at release from manufacturing (by Day 0 [infusion day] for each participant)
  No more than two products fail the target cell dose and established release criteria.
Find the safe maximum tolerated dose | Up to 60 days post-infusion for each participant
  No more than 1 out of 6 participants may experience a related dose limiting toxicity or treatment emergent adverse events.

SECONDARY OUTCOMES:
Change in Diarrhea incidence | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (daily for the first month followed by monthly at Month 2, 3, 6, 9, 12)
  Stool Diary records - extent of diarrhea as measured by frequency and volume of stools, and the presence or absence of blood and/or mucus, and stool studies at specified time points (for all ages).
Change in GI Symptoms - Gastrointestinal Symptoms Rating Scale | Baseline (up to 60 days before infusion of CD4^LVFOXP3) through post-infusion (Week 4, Month 6, Month 12)
  Gastrointestinal Symptoms Rating Scale (GSRS) (for patients ≥12 years old).
Change in Body Mass Index (BMI) | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 1, 2, 3, Week 1, 2, 3, 4; Month 2, 3, 6, 9, 12)
  BMI measured as kg/m^2.
Change in age-specific percentiles of height | Baseline (up to 60 days before infusion of CD4^LVFOXP3) through post-infusion (Month 12)
Change in age-specific percentiles of bodyweight | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 1, 2, 3, Week 1, 2, 3, 4; Month 2, 3, 6, 9, 12)
Change in Bilirubin levels | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 2, Week 1, 2, 3, 4; Month 2, 3, 6, 9 and 12)
Change in Liver Enzyme - Alanine Transaminase (ALT) | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 2, Week 1, 2, 3, 4; Month 2, 3, 6, 9 and 12)
Change in Liver Enzyme - Aspartate Transaminase (AST) | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 2, Week 1, 2, 3, 4; Month 2, 3, 6, 9 and 12)
Change in Liver Enzyme - Alkaline Phosphatase (ALP) | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 2, Week 1, 2, 3, 4; Month 2, 3, 6, 9 and 12)
Change in Liver Enzyme - Gamma Glutyltranspeptidase (GGT) | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 2, Week 1, 2, 3, 4; Month 2, 3, 6, 9 and 12)
Change in INR level | Baseline/screening (up to 60 days before infusion of CD4^LVFOXP3) through post-infusion (Week 4; Month 3, 6, 12)
  International normalized ratio (INR) to determine prothrombin time.
Skin Disease (EASI) - Changes from Baseline/ Pre-infusion | Baseline (up to 60 days before infusion of CD4^LVFOXP3), through post-infusion (Day 1; Week 1, 2, 3, 4; Month 3, 6 and 12)
  Scoring of areas of involvement in each anatomical region (area), calculation of intensity using Eczema Area and Severity Index (EASI).
Skin Disease (POEM) - Changes from Baseline/ Pre-infusion | Baseline (up to 60 days before infusion of CD4^LVFOXP3), through post-infusion (Day 1; Week 1, 2, 3, 4; Month 3, 6 and 12)
  Scoring of areas of involvement in each anatomical region (area), calculation of intensity using Patient oriented eczema measure (POEM).
Skin Disease (PASI) - Changes from Baseline/ Pre-infusion | Baseline (up to 60 days before infusion of CD4^LVFOXP3), through post-infusion (Day 1; Week 1, 2, 3, 4; Month 3, 6 and 12)
  Changes in the extent (%) and severity of skin lesions and their complications (i.e. infections, atrophy, itching) using Psoriasis Area and Severity Index (PASI).
Skin Disease (MTLSS) - Changes from Baseline/ Pre-infusion | Baseline (up to 60 days before infusion of CD4^LVFOXP3), through post-infusion (Day 1; Week 1, 2, 3, 4; Month 3, 6 and 12)
  Changes in the extent (%) and severity of skin lesions and their complications (i.e. infections, atrophy, itching) using Modified Total Lesional Sign Score (MTLSS).
Change in skin barrier function | Baseline (up to 60 days before infusion of CD4^LVFOXP3), through post-infusion (Day 1; Week 1, 2, 3, 4; Month 3, 6 and 12)
  Biophysical Skin Evaluation: Skin measurement of transepidermal water loss to monitor skin barrier function and erythema
Change in Hemolytic Anemia (RBC) | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 1, 2, 3; Week 1, 2, 3, 4; Month 2, 3, 6, 9, 12)
  Measurement of the number of red blood cells (Complete Blood Counts with Differential [CBCD]).
Change in Hemolytic Anemia (Reticulocyte) | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 1, 2, 3; Week 1, 2, 3, 4; Month 2, 3, 6, 9, 12)
  Measurement of the number of reticulocytes.
Change in Thrombocytopenia | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 1, 2, 3; Week 1, 2, 3, 4; Month 2, 3, 6, 9, 12)
  Measure the number of platelets (Complete Blood Counts with Differential (CBCD)).
Change in Neutropenia | Baseline (up to 60 days before infusion of CD4^LVFOXP3), pre-infusion through post-infusion (Day 1, 2, 3; Week 1, 2, 3, 4; Month 2, 3, 6, 9, 12)
  Measure the number of neutrophils (Complete Blood Counts with Differential [CBCD]).
Change in C-peptide - Type 1 diabetes Pre-onset | Baseline taken 60-30 days before infusion of CD4^LVFOXP3; Post-infusion (Week 4, Month 3, 6 and 12).
Change in HbA1c - Type 1 diabetes Pre-onset | Baseline taken 60-30 days before infusion of CD4^LVFOXP3; Post-infusion (Week 4, Month 3, 6 and 12).
Change in Daily insulin requirement - Type 1 diabetes monitoring | Baseline taken 60-30 days before infusion of CD4^LVFOXP3 and post-infusion (over 7 consecutive days preceding each study visit);
  Mean daily insulin use recorded over 7 consecutive days preceding each evaluation timepoint for patients with Type 1 Diabetes.
Change in hyper-/hypo-glycemic events - Type 1 diabetes monitoring | Baseline taken 60-30 days before infusion of CD4^LVFOXP3 and post-infusion (over 7 consecutive days preceding each study visit);
  Continuous glucose monitoring (CGM) metrics to log episodes of hyper/hypoglycemic events.
Change in Autoantibody Profile | Screening/ Baseline, Post-infusion (Month 6 and 12)
  Measure autoantibodies to organs involved in the disease (participant-specific): anti-insulin (IAA), anti-islet antigens (IA), anti-glutamic acid decarboxylase (GAD), anti-zinc transporter8 (ZNT8), anti-islet cells (ICA), anti-liver kidney microsome (LKM), anti-thyroperoxidase (TPO), anti-thyroglobulin (TG), anti-enterocytes, anti-SMA
Change in Creatinine as a measure of Kidney Function | Baseline taken 60-30 days before infusion of CD4^LVFOXP3, Pre-infusion, Week 1, 2, 3, 4; Month 2, 3, 6, 9 and 12
  Measure kidney functional parameters, i.e., creatinine, in the blood and urine.
Change in PedsQL General Well-Being Scale - Quality of Life | Pre-Infusion; Month 6, 12
Change in PedsQL Generic Core Scale - Quality of Life | Pre-Infusion; Month 6, 12
Change in PedsQL Gastrointestinal Symptoms Scale - Quality of Life | Pre-Infusion; Month 6, 12
  Measured with Gastrointestinal Symptoms Scale: minimum value = 0 (never a problem), maximum value = 4 (almost always a problem). Higher scores mean a worse outcome.
Disease-free Survival - Changes from Baseline | Up to 15 years
  The length of time from cell infusion to the point at which the participant survives without any new or worsening of existing signs or symptoms of disease. The data will be compared with historical disease-free survival probability. Probability of disease-free survival will be computed with the use of Kaplan-Meier estimator.
Overall Survival - Changes from Baseline | Up to 15 years
  Participant survival

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Alexander, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allan SE, Alstad AN, Merindol N, Crellin NK, Amendola M, Bacchetta R, Naldini L, Roncarolo MG, Soudeyns H, Levings MK. Generation of potent and stable human CD4+ T regulatory cells by activation-independent expression of FOXP3. Mol Ther. 2008 Jan;16(1):194-202. doi: 10.1038/sj.mt.6300341. Epub 2007 Nov 6. PMID 17984976
- [Background] Amendola M, Venneri MA, Biffi A, Vigna E, Naldini L. Coordinate dual-gene transgenesis by lentiviral vectors carrying synthetic bidirectional promoters. Nat Biotechnol. 2005 Jan;23(1):108-16. doi: 10.1038/nbt1049. Epub 2004 Dec 26. PMID 15619618
- [Background] Baecher-Allan CM, Hafler DA. The purification and functional analysis of human CD4+CD25high regulatory T cells. Curr Protoc Immunol. 2006 May;Chapter 7:7.4B.1-7.4B.12. doi: 10.1002/0471142735.im0704bs72. PMID 18432975
- [Background] Barzaghi F, Passerini L, Gambineri E, Ciullini Mannurita S, Cornu T, Kang ES, Choe YH, Cancrini C, Corrente S, Ciccocioppo R, Cecconi M, Zuin G, Discepolo V, Sartirana C, Schmidtko J, Ikinciogullari A, Ambrosi A, Roncarolo MG, Olek S, Bacchetta R. Demethylation analysis of the FOXP3 locus shows quantitative defects of regulatory T cells in IPEX-like syndrome. J Autoimmun. 2012 Feb;38(1):49-58. doi: 10.1016/j.jaut.2011.12.009. Epub 2012 Jan 20. PMID 22264504
- [Background] Barzaghi F, Amaya Hernandez LC, Neven B, Ricci S, Kucuk ZY, Bleesing JJ, Nademi Z, Slatter MA, Ulloa ER, Shcherbina A, Roppelt A, Worth A, Silva J, Aiuti A, Murguia-Favela L, Speckmann C, Carneiro-Sampaio M, Fernandes JF, Baris S, Ozen A, Karakoc-Aydiner E, Kiykim A, Schulz A, Steinmann S, Notarangelo LD, Gambineri E, Lionetti P, Shearer WT, Forbes LR, Martinez C, Moshous D, Blanche S, Fisher A, Ruemmele FM, Tissandier C, Ouachee-Chardin M, Rieux-Laucat F, Cavazzana M, Qasim W, Lucarelli B, Albert MH, Kobayashi I, Alonso L, Diaz De Heredia C, Kanegane H, Lawitschka A, Seo JJ, Gonzalez-Vicent M, Diaz MA, Goyal RK, Sauer MG, Yesilipek A, Kim M, Yilmaz-Demirdag Y, Bhatia M, Khlevner J, Richmond Padilla EJ, Martino S, Montin D, Neth O, Molinos-Quintana A, Valverde-Fernandez J, Broides A, Pinsk V, Ballauf A, Haerynck F, Bordon V, Dhooge C, Garcia-Lloret ML, Bredius RG, Kalwak K, Haddad E, Seidel MG, Duckers G, Pai SY, Dvorak CC, Ehl S, Locatelli F, Goldman F, Gennery AR, Cowan MJ, Roncarolo MG, Bacchetta R; Primary Immune Deficiency Treatment Consortium (PIDTC) and the Inborn Errors Working Party (IEWP) of the European Society for Blood and Marrow Transplantation (EBMT). Long-term follow-up of IPEX syndrome patients after different therapeutic strategies: An international multicenter retrospective study. J Allergy Clin Immunol. 2018 Mar;141(3):1036-1049.e5. doi: 10.1016/j.jaci.2017.10.041. Epub 2017 Dec 11. PMID 29241729
- [Background] Battaglia M, Stabilini A, Roncarolo MG. Rapamycin selectively expands CD4+CD25+FoxP3+ regulatory T cells. Blood. 2005 Jun 15;105(12):4743-8. doi: 10.1182/blood-2004-10-3932. Epub 2005 Mar 3. PMID 15746082
- [Background] Bluestone JA, Tang Q. Treg cells-the next frontier of cell therapy. Science. 2018 Oct 12;362(6411):154-155. doi: 10.1126/science.aau2688. No abstract available. PMID 30309932
- [Background] Bluestone JA, Buckner JH, Fitch M, Gitelman SE, Gupta S, Hellerstein MK, Herold KC, Lares A, Lee MR, Li K, Liu W, Long SA, Masiello LM, Nguyen V, Putnam AL, Rieck M, Sayre PH, Tang Q. Type 1 diabetes immunotherapy using polyclonal regulatory T cells. Sci Transl Med. 2015 Nov 25;7(315):315ra189. doi: 10.1126/scitranslmed.aad4134. PMID 26606968
- [Background] Bonini C, Grez M, Traversari C, Ciceri F, Marktel S, Ferrari G, Dinauer M, Sadat M, Aiuti A, Deola S, Radrizzani M, Hagenbeek A, Apperley J, Ebeling S, Martens A, Kolb HJ, Weber M, Lotti F, Grande A, Weissinger E, Bueren JA, Lamana M, Falkenburg JH, Heemskerk MH, Austin T, Kornblau S, Marini F, Benati C, Magnani Z, Cazzaniga S, Toma S, Gallo-Stampino C, Introna M, Slavin S, Greenberg PD, Bregni M, Mavilio F, Bordignon C. Safety of retroviral gene marking with a truncated NGF receptor. Nat Med. 2003 Apr;9(4):367-9. doi: 10.1038/nm0403-367. No abstract available. PMID 12669036
- [Background] Brunkow ME, Jeffery EW, Hjerrild KA, Paeper B, Clark LB, Yasayko SA, Wilkinson JE, Galas D, Ziegler SF, Ramsdell F. Disruption of a new forkhead/winged-helix protein, scurfin, results in the fatal lymphoproliferative disorder of the scurfy mouse. Nat Genet. 2001 Jan;27(1):68-73. doi: 10.1038/83784. PMID 11138001
- [Background] Consonni F, Ciullini Mannurita S, Gambineri E. Atypical Presentations of IPEX: Expect the Unexpected. Front Pediatr. 2021 Feb 5;9:643094. doi: 10.3389/fped.2021.643094. eCollection 2021. PMID 33614561
- [Background] Brunstein CG, Miller JS, McKenna DH, Hippen KL, DeFor TE, Sumstad D, Curtsinger J, Verneris MR, MacMillan ML, Levine BL, Riley JL, June CH, Le C, Weisdorf DJ, McGlave PB, Blazar BR, Wagner JE. Umbilical cord blood-derived T regulatory cells to prevent GVHD: kinetics, toxicity profile, and clinical effect. Blood. 2016 Feb 25;127(8):1044-51. doi: 10.1182/blood-2015-06-653667. Epub 2015 Nov 12. PMID 26563133
- [Background] Cornetta K, Duffy L, Turtle CJ, Jensen M, Forman S, Binder-Scholl G, Fry T, Chew A, Maloney DG, June CH. Absence of Replication-Competent Lentivirus in the Clinic: Analysis of Infused T Cell Products. Mol Ther. 2018 Jan 3;26(1):280-288. doi: 10.1016/j.ymthe.2017.09.008. Epub 2017 Sep 12. PMID 28970045
- [Background] Delville M, Bellier F, Leon J, Klifa R, Lizot S, Vincon H, Sobrino S, Thouenon R, Marchal A, Garrigue A, Olivre J, Charbonnier S, Lagresle-Peyrou C, Amendola M, Schambach A, Gross D, Lamarthee B, Benoist C, Zuber J, Andre I, Cavazzana M, Six E. A combination of cyclophosphamide and interleukin-2 allows CD4+ T cells converted to Tregs to control scurfy syndrome. Blood. 2021 Apr 29;137(17):2326-2336. doi: 10.1182/blood.2020009187. PMID 33545713
- [Background] Fontenot JD, Gavin MA, Rudensky AY. Foxp3 programs the development and function of CD4+CD25+ regulatory T cells. Nat Immunol. 2003 Apr;4(4):330-6. doi: 10.1038/ni904. Epub 2003 Mar 3. PMID 12612578
- [Background] Gambineri E, Perroni L, Passerini L, Bianchi L, Doglioni C, Meschi F, Bonfanti R, Sznajer Y, Tommasini A, Lawitschka A, Junker A, Dunstheimer D, Heidemann PH, Cazzola G, Cipolli M, Friedrich W, Janic D, Azzi N, Richmond E, Vignola S, Barabino A, Chiumello G, Azzari C, Roncarolo MG, Bacchetta R. Clinical and molecular profile of a new series of patients with immune dysregulation, polyendocrinopathy, enteropathy, X-linked syndrome: inconsistent correlation between forkhead box protein 3 expression and disease severity. J Allergy Clin Immunol. 2008 Dec;122(6):1105-1112.e1. doi: 10.1016/j.jaci.2008.09.027. Epub 2008 Oct 25. PMID 18951619
- [Background] Gambineri E, Ciullini Mannurita S, Hagin D, Vignoli M, Anover-Sombke S, DeBoer S, Segundo GRS, Allenspach EJ, Favre C, Ochs HD, Torgerson TR. Clinical, Immunological, and Molecular Heterogeneity of 173 Patients With the Phenotype of Immune Dysregulation, Polyendocrinopathy, Enteropathy, X-Linked (IPEX) Syndrome. Front Immunol. 2018 Nov 1;9:2411. doi: 10.3389/fimmu.2018.02411. eCollection 2018. PMID 30443250
- [Background] Hori S, Nomura T, Sakaguchi S. Control of regulatory T cell development by the transcription factor Foxp3. Science. 2003 Feb 14;299(5609):1057-61. doi: 10.1126/science.1079490. Epub 2003 Jan 9. PMID 12522256
- [Background] Marek-Trzonkowska N, Mysliwiec M, Dobyszuk A, Grabowska M, Derkowska I, Juscinska J, Owczuk R, Szadkowska A, Witkowski P, Mlynarski W, Jarosz-Chobot P, Bossowski A, Siebert J, Trzonkowski P. Therapy of type 1 diabetes with CD4(+)CD25(high)CD127-regulatory T cells prolongs survival of pancreatic islets - results of one year follow-up. Clin Immunol. 2014 Jul;153(1):23-30. doi: 10.1016/j.clim.2014.03.016. Epub 2014 Apr 1. PMID 24704576
- [Background] Passerini L, Rossi Mel E, Sartirana C, Fousteri G, Bondanza A, Naldini L, Roncarolo MG, Bacchetta R. CD4(+) T cells from IPEX patients convert into functional and stable regulatory T cells by FOXP3 gene transfer. Sci Transl Med. 2013 Dec 11;5(215):215ra174. doi: 10.1126/scitranslmed.3007320. PMID 24337481
- [Background] Passerini L, Barzaghi F, Curto R, Sartirana C, Barera G, Tucci F, Albarello L, Mariani A, Testoni PA, Bazzigaluppi E, Bosi E, Lampasona V, Neth O, Zama D, Hoenig M, Schulz A, Seidel MG, Rabbone I, Olek S, Roncarolo MG, Cicalese MP, Aiuti A, Bacchetta R. Treatment with rapamycin can restore regulatory T-cell function in IPEX patients. J Allergy Clin Immunol. 2020 Apr;145(4):1262-1271.e13. doi: 10.1016/j.jaci.2019.11.043. Epub 2019 Dec 23. PMID 31874182
- [Background] Sakaguchi S, Sakaguchi N, Asano M, Itoh M, Toda M. Immunologic self-tolerance maintained by activated T cells expressing IL-2 receptor alpha-chains (CD25). Breakdown of a single mechanism of self-tolerance causes various autoimmune diseases. J Immunol. 1995 Aug 1;155(3):1151-64. PMID 7636184
- [Background] Sato Y, Passerini L, Piening BD, Uyeda MJ, Goodwin M, Gregori S, Snyder MP, Bertaina A, Roncarolo MG, Bacchetta R. Human-engineered Treg-like cells suppress FOXP3-deficient T cells but preserve adaptive immune responses in vivo. Clin Transl Immunology. 2020 Nov 25;9(11):e1214. doi: 10.1002/cti2.1214. eCollection 2020. PMID 33304583